CLINICAL TRIAL: NCT06803069
Title: Investigation of the Mechanisms of the Tendency to Hypothermia in Newborns and Premature Infants During Surgical Interventions and in the Intensive Care Unit (Non-Interventional, Single-Center, Prospective Clinical Research)
Brief Title: Investigation of the Mechanisms of the Tendency to Hypothermia in Newborns and Premature Neonates
Status: Recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: BM/17552-3/2024; NKFIH-FK-138722 (Other Grant/Funding Number: National Research, Development and Innovation Office)
Record Dates: First submitted 2025-01-25; First posted 2025-01-31 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Hypothermia; Brown Adipose Tissue; Preterm and Term Infants; Neonate; Thermogenesis; Blood Markers
Keywords: brown adipose tissue; neonate; neonatal hypothermia; preterm; nonshivering thermogenesis; infant; newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preterm neonates: Group of neonates who were born before the 37th gestational week.
- Full-term neonates: Group of neonates who were born after the 37th gestational week.

SUMMARY:
Newborns have thermoregulatory mechanisms that differ from those of adults. Instead of producing heat through shivering, newborns primarily rely on non-shivering thermogenesis by the brown adipose tissue. The development of this thermogenic tissue starts around the 26th gestational week and continues until shortly before birth, after which no further growth occurs. As a result, premature infants, who have less developed brown fat, are more prone to reduced heat production and are at higher risk for hypothermia. There are few human studies examining the thermoregulatory differences and mechanisms between full-term and premature neonates, and the findings remain inconclusive.

In this study, the investigators aim to conduct a prospective, observational research. Researchers will compare body temperature, brown adipose tissue activity, and specific plasma markers between full-term and premature neonates in insensive care units and during elective surgeries.

DETAILED DESCRIPTION:
Test Methods:

Both substudies involve the use of a FLIR C3 mobile thermal camera to create thermograms. Thermal images of the full-term and preterm infants are taken from a distance of 20 cm while the participants lie in a supine position. The area examined spans from the upper edge of the diaper to the top of the head.

Substudy 1:

1. a) In case of neonates in the intensive care unit or waiting for short procedures (e.g., ophthalmic surgery), thermal images are taken before transport to the operating room and after surgery, before transferring back to the ward. For infants receiving incubator care, both images are taken inside the transport incubator. The test duration is about 5 minutes.

1. b) Images are captured before kangaroo care, before and after transferring the infant to the ward (both images taken in the transport incubator if the infant is in incubator care).

1. c) Thermal images are taken before and after the insertion of an epicutaneous cannula.

1. d) For post-asphyxic infants undergoing therapeutic hypothermia, images are taken immediately before starting cooling on the therapeutic mattress, once midway through the cooling process; once immediately after reaching the target core temperature; then daily while in the hypothermic state; once immediately before the rewarming process, and every hour during rewarming until the desired core temperature is reached.

   Substudy 2:
2. a) In case of neonates waiting for surgeries lasting more than 30 minutes, thermal images are taken before the surgery; every 10 minutes during the operation; after surgery, following the same protocol as in Substudy 1.

2. b) Thermal images are taken before and after inserting a central cannula.

Parameters recorded in the substudies:

1. Blood tests, including c-reactive protein (CRP), procalcitonin (PCT), blood count, glucose, bilirubin, thyroid hormones, urea, creatinine, glutamate oxaloacetate transaminase (GOT), glutamate pyruvate transaminase (GPT), lactate dehydrogenase (LDH), gamma-glutamyl transferase (GGT), and blood gas, as part of routine blood sampling.
2. Rectal core temperature, as well as episodes of shivering or heat production.
3. Changes in body temperature during surgery along with other routinely measured physiological parameters (e.g., blood pressure, respiratory indicators).
4. Type and dosage of anesthetics used, as well as any side effects (e.g., post-surgery vomiting).
5. Additional parameters such as gestational age, Apgar score, birth weight, body weight at the time of examination, and environmental temperature (e.g., clinic, incubator, operating room).

Examination process:

The parents/guardians/legal representatives of the selected patients will be provided with detailed information, and consent forms will be signed by them.

ELIGIBILITY:
Inclusion Criteria:

* For Substudy 1: Patients admitted to the Neonatal Intensive Care Unit at the University of Pécs, Department of Obstetrics and Gynaecology (premature infants or those in neonatal intensive care).
* For Substudy 2: Patients under 2 years of age undergoing elective surgery lasting more than 30 minutes at the University of Pécs, Department of Paediatrics.
* For both substudies: Written consent for participation in the study has been provided by the patient's parent, guardian, or legal representative.

Exclusion Criteria:

* For both substudies: If the patient cannot be mobilized (e.g., during the post-operative phase of abdominal or thoracic surgery; presence of chest tubes for pneumothorax or other reasons; hemodynamic instability; need for continuous electrocardiogram (ECG) monitoring; or use of an external pacemaker).
* The patient's parent, guardian, or legal representative does not consent to the study or withdraws their consent at any point.
* For Substudy 2: if the patient is older than 2 years.

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population consist of randomly chosen preterm and full-term neonates.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Temperature data from the back of neonates revealing brown adipose tissue activity | 2 years
  Primary objective (Primary endpoint):
  The thermogram analysis may reveal reduced brown adipose tissue activity in preterm infants, which could contribute to their increased susceptibility to hypothermia during surgeries and intensive care. The temperature values of the head, brown fat, and trunk will be recorded in degrees of Celsius (°C) with thermal imaging. Their difference (e.g., brown fat temperature minus trunk temperature) will be used as a measure of brown fat activity also expressed in °C.

SECONDARY OUTCOMES:
Concentration and count of special laboratory parameters in connection with thermogenesis in neonates | 3 years
  Secondary objective (Secondary endpoint):
  Blood test parameters of the newborns will be determined by the accredited Medical Testing Laboratory at the Clinical Centre, University of Pecs. These include blood cell counts [red blood cells (T/l), white blood cells (G/l), and platelets (G/l)], hemoglobin (g/l), hematocrit (%), glucose (mmol/l), bilirubin (µmol/l), thyroid hormones (mIU/l), urea (µmol/l), creatinine (µmol/l), CRP (mg/l), AST (IU/l), ALT (IU/l), GGT (IU/l), LDH (IU/l), PCT (0,5 ng/ml). They will be used to assess correlations between brown fat activity (see Primary Outcome Measure) and blood levels of a given blood parameter.
Blood cell counts | 3 years
  Level of red blood cells in T/l, white blood cells in G/l, and platelets in G/l.
Hemoglobin level | 3 years
  Hemoglobin level in g/l
Hematocrit level | 3 years
  Hematocrit level in %.
Glucose level | 3 years
  Glucose level in mmol/l.
Liver fuction | 3 years
  bilirubin in µmol/l, AST in IU/l, ALT in IU/l, GGT in IU/l, LDH in IU/l.
Kidney function | 3 years
  urea in µmol/l, creatinine in µmol/l.
Thyroid function | 3 years
  thyroid hormones in mIU/l (TSH, T3, T4).
Inflammatory markers | 3 years
  CRP in mg/l and PCT in ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Tamás Kövesi, MD, PhD, Principal Investigator — University of Pecs, Department of Anaesthesiology and Intensive Therapy; András Garami, MD, PhD, Principal Investigator — University of Pecs, Institute for Translational Medicine; Simone Funke, MD, PhD, Principal Investigator — University of Pecs, Department of Obstetrics and Gynaecology
Locations (2):
- Hungary (2):
  - University of Pécs, Department of Obstetrics and Gynaecology, Pécs, Baranya
  - University of Pécs, Department of Paediatrics, Pécs, Baranya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nedergaard J, Cannon B. Brown adipose tissue as a heat-producing thermoeffector. Handb Clin Neurol. 2018;156:137-152. doi: 10.1016/B978-0-444-63912-7.00009-6. PMID 30454587
- [Background] Symonds ME, Pope M, Sharkey D, Budge H. Adipose tissue and fetal programming. Diabetologia. 2012 Jun;55(6):1597-606. doi: 10.1007/s00125-012-2505-5. Epub 2012 Mar 9. PMID 22402988
- [Background] Lunze K, Hamer DH. Thermal protection of the newborn in resource-limited environments. J Perinatol. 2012 May;32(5):317-24. doi: 10.1038/jp.2012.11. Epub 2012 Mar 1. PMID 22382859
- [Background] Silverman WA, Sinclair JC. Temperature regulation in the newborn infant. N Engl J Med. 1966 Jan 13;274(2):92-4 contd. doi: 10.1056/NEJM196601132740207. No abstract available. PMID 5322157
- [Background] Knobel R, Holditch-Davis D. Thermoregulation and heat loss prevention after birth and during neonatal intensive-care unit stabilization of extremely low-birthweight infants. J Obstet Gynecol Neonatal Nurs. 2007 May-Jun;36(3):280-7. doi: 10.1111/j.1552-6909.2007.00149.x. PMID 17489935
- [Background] Lidell ME. Brown Adipose Tissue in Human Infants. Handb Exp Pharmacol. 2019;251:107-123. doi: 10.1007/164_2018_118. PMID 29675580